CLINICAL TRIAL: NCT05956418
Title: A Prospective, Multi-centric, Open-labeled, Phase-IV Study to Assess Safety and Efficacy of LYFAQUIN™ (Centhaquine Citrate) as a Resuscitative Agent for Hypovolemic Shock to be Used as an Adjuvant to Standard Treatment of Shock
Brief Title: A Study to Assess the Safety and Efficacy of Centhaquine in Hypovolemic Shock Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmazz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMZ-2010/CT-4.1/2019
Record Dates: First submitted 2023-06-30; First posted 2023-07-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hypovolemic Shock
Keywords: Shock; Hypovolemia; Hemorrhage; Blood Pressure; Resuscitation; Centhaquine; Adrenergic
MeSH Terms: conditions — Shock; Hypovolemia; Hemorrhage | interventions — centhaquine

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-centric, open-labeled, single-arm and phase-IV study in 400 hypovolemic shock patients with a systolic arterial blood pressure ≤ 90 mmHg. The study duration will be approximately 15 months, including a 12-month enrollment period. All patients in the single group of the study will receive treatment with "Centhaquine (Dose: 0.01 mg/kg) + Standard of care." A second dose of centhaquine may be given if the systolic blood pressure remains low. However, the maximum number of doses per day should not exceed 3, and if needed the treatment will continue for the 2nd day of enrollment. Within the first 48 hours post-enrollment, a minimum of 1 dose and a maximum of 6 doses of centhaquine will be administered. Each patient will be closely monitored throughout their hospitalization and followed until discharge or day 7 (whichever comes earlier) from enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Centhaquine (Dose: 0.01 mg/kg) + Standard of care (Experimental): Centhaquine will be administered intravenously after enrollment to hypovolemic shock patients with systolic arterial blood pressure ≤ 90 mmHg at presentation and continue to receive standard shock treatment. Centhaquine will be administered at a dose of 0.01 mg/kg of body weight, as an intravenous (IV) infusion over 1 hour in 100 mL of normal saline. Second dose of centhaquine will be administered if SBP falls below or remains below or equal to 90 mmHg but not before 4 hours of the previous dose and total doses per day (in 24 hours) will not exceed 3 doses. Centhaquine administration if needed will continue for two days post-enrollment. A minimum of 1 dose or maximum of 6 doses of centhaquine will be administered within first 48 hours post-enrollment. Each patient will be monitored closely throughout his/her hospitalization and will be followed until discharge or day 7 (whichever is earlier) from enrollment.
  Interventions: Drug: Centhaquine

INTERVENTIONS:
Drug: Centhaquine — Centhaquine (LYFAQUIN™ or centhaquine citrate) is a novel, first-in-class, highly effective resuscitative agent for hypovolemic shock. Phase II results demonstrate highly significant efficacy in improving blood pressure (p<0.0001), lactate levels (p=0.0012) and base-deficit (p<0.0001). There was also improvement in reduction in use of vasopressors and reduced mortality. Similarly, results of phase III study confirmed the safety and efficacy of centhaquine as an adjuvant to standard of care for hypovolemic shock. Therefore, to assess safety of centhaquine in large population a phase IV study (post-authorization safety study) has been designed.
  Other Names: LYFAQUIN™; Centhaquine Citrate; 2-(2-(4-(3-methylphenyl)-1-piperazinyl)ethyl) quinoline citrate; PMZ-2010

SUMMARY:
This is a prospective, multi-centric, open-labeled, phase-IV clinical study to evaluate the safety and efficacy of centhaquine citrate (LYFAQUIN™), a first-in-class drug for treating hypovolemic shock, a life-threatening condition caused by severe blood or fluid loss. Centhaquine has been found to be an effective resuscitative agent in rat, rabbit, and swine models of hemorrhagic shock. It has demonstrated the ability to decrease blood lactate levels, increase mean arterial pressure, enhance cardiac output, and reduce mortality rates. The increase in cardiac output during resuscitation is primarily attributed to an augmentation in stroke volume. Centhaquine exerts its effects by acting on the venous α2B-adrenergic receptors, which enhances venous return to the heart. Additionally, it produces arterial dilation by targeting central α2A-adrenergic receptors, thereby reducing sympathetic activity and systemic vascular resistance.

DETAILED DESCRIPTION:
This study will enroll approximately 400 patients aged 18 years or older with hypovolemic shock and a systolic blood pressure of 90 mmHg or lower upon admission to the hospital. These patients will continue to receive standard shock treatment, including endotracheal intubation, fluid resuscitation, and vasopressors. The trial seeks to answer several key questions: Is centhaquine safe to use in patients with hypovolemic shock? Can centhaquine improve blood pressure, lactate levels, and base deficit, and reduce mortality? Participants will receive centhaquine in addition to the standard of care. Centhaquine will be administered intravenously in 100 mL of normal saline at a dose of 0.01 mg/kg of body weight over a period of one hour. A second dose will be given if the systolic blood pressure remains at or below 90 mmHg, but not before 4 hours have passed since the previous dose. The total number of doses within 24 hours will not exceed 3, and centhaquine administration may continue for up to two days after enrollment. Each patient will be closely monitored throughout their hospitalization and followed until discharge or up to seven days from enrollment, whichever comes first. The trial will assess safety and efficacy parameters according to a predefined schedule of visits. The baseline characteristics of the patients in different groups will be compared using statistical tests such as the Chi-square test for categorical variables and the Unpaired t-test for continuous variables. Changes in dichotomous variables between groups from baseline to follow-ups will be analyzed using McNemar's test. Survival rates will be measured using Kaplan-Meier survival analysis, and univariate and multiple Cox-regression analysis will be employed to determine hazard ratios and their 95% confidence intervals for patient survival. The trial results will be presented as mean±SEM (median, minimum, and maximum) values and percentages.

ELIGIBILITY:
Inclusion Criteria

• Adult hypovolemic shock patients aged 18 years or older admitted to the emergency room or ICU with systolic blood pressure ≤ 90 mmHg at presentation and continue to receive standard shock treatment. Blood Lactate level indicative of hypovolemic shock (>2.0 mmol/L).

Exclusion Criteria

* Development of any other terminal illness not associated with hypovolemic shock during the study duration.
* Patient with altered consciousness not due to hypovolemic shock and comatose patient. • Known pregnancy.
* Cardiopulmonary resuscitation (CPR) before enrollment.
* Presence of a do not resuscitate order.
* Patient is participating in another interventional study.
* Patients with systemic diseases which were already present before having trauma, such as sepsis, cancer, chronic renal failure, liver failure, decompensated heart failure, or AIDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with adverse events (AEs) and serious adverse events (SAEs) | Up to 7 days
  Any unfavorable sign, symptom, or disease that occurs while using centhaquine will be reported as an adverse event (AE), including worsening of pre-existing medical conditions. A severe medical occurrence, such as death, life-threatening situations, hospitalization, significant disability, or congenital anomalies will be reported as a serious adverse event (SAE). AEs will be collected through patient questioning, spontaneous reports, and observation. Description, severity, start and end dates, incidence, relationship to the centhaquine, seriousness, action taken, and outcome of AEs will be documented in source documents and case report forms (CRFs). All SAEs will be reported within 24 hours to the sponsor, Drugs Controller General of India, and the ethics committee. Follow-up information and hospitalization or autopsy reports will be provided if necessary. A detailed analyzed report of all SAEs will be prepared and submitted to relevant authorities within 14 days.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | Up to 7 days
  Hypovolemia is known to cause low blood pressure, severely. That may lead to multi-organ failure or death. Hence, improving blood pressure is the key to the development of effective hypovolemic shock therapeutics.
Blood lactate | 48 hours
  Increased blood lactate level is indicative of hypovolemic shock. Lactate level of more than 2 mmol/L is correlated with increased tissue hypoxia and anaerobic respiration following shock.
Base-deficit | 48 hours
  The base deficit is a known measure of metabolic acidosis and has been advocated as a marker of resuscitation adequacy. It is correlated with the severity of injury and degree of hemorrhage, which makes it useful in the operating room (OR) as an endpoint of resuscitation.
Time in intensive care unit (ICU) | Up to 7 days
  In the intensive care unit, specific medical specialties will be provided to support the shock patients whose lives are in immediate danger. ICU medical interventions take over the function of defective or damaged organs and maintain blood pressure in shock patients.
Time on ventilator | Up to 7 days
  Ventilatory support is commonly used to resolve the circulation problem in shock patients.
Urine output | 48 hours
  The urine output is an important clinical parameter for renal function and blood volume status, especially in critically ill multiple trauma patients during their hospital admission and ICU. Also, it is a reliable incipient marker of hypovolemia therefore it has a place among the parameters used to monitor the hemodynamic status of critically ill multiple trauma patients.
Incidence of mortality | 7 days
  The hypovolemic shock causes ischemic injury to vital organs and may lead to multi-system organ failure and death (mortality).
Multiple Organ Dysfunction Syndrome score (MODS) | Up to 7 days
  Multiple organ dysfunction syndrome (MODS) is a life-threatening complication and a major cause of mortality in the injured patient. MODS is a 5-grade scale from 0 to 4, where 0 is the best and 4 is the worst outcome.
Acute Respiratory Distress Syndrome (ARDS) | Up to 7 days
  Acute respiratory distress syndrome (ARDS) is a serious lung condition, which causes low blood oxygen. It is a complication of shock associated with hypovolemia, hypoxemia, and inadequate cardiovascular compensatory responses to increased O2 demands. It is preceded by hypovolemia, reduced heart function, inadequate O2 delivery, and extraction needed to maintain VO2 in injured patients with increased metabolic as well as O2 requirements.
Glasgow Coma Scale (GCS) | Up to 7 days
  Glasgow Coma Scale (GCS) is a neurological scale consisting of the sum of three coded values: motor, verbal, and eye-opening. It provides a reliable way of recording the conscious state of a person or shock patient. GCS is a 15-point scale to assess the level of consciousness of patients where less than 3 is a comatose state and 15 is fully awake.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Lavhale, Ph.D., Study Director — Pharmazz India
Locations (17):
- India (17):
  - ACSR Government Medical College and Hospital, Nellore, Andhra Pradesh
  - All India Institute of Medical Sciences (AIIMS), Raipur, Chhattisgarh
  - Aman Hospital, Vadodara, Gujarat
  - New Era Hospital, Nagpur, Maharashtra
  - Seven Star Hospital, Nagpur, Maharashtra
  - Meditrina Hospital, Nagpur, Maharashtra
  - Sri Guru Ram Das University of Health Sciences (SGRDH), Amritsar, Punjab
  - Dayanand Medical College & Hospital (DMCH), Ludhiana, Punjab
  - Christian Medical College and Hospital (CMC), Ludhiana, Punjab
  - Government Medical College, Kota, Rajasthan
  - KG Hospital, Coimbatore, Tamil Nadu
  - Pushpanjali Hospital, Agra, Uttar Pradesh
  - Maharani Laxmi Bai Medical College (MLBMC), Jhānsi, Uttar Pradesh
  - Nirmal Hospital, Jhānsi, Uttar Pradesh
  - Ganesh Shankar Vidyarthi Memorial Medical College (GSVM), Kanpur, Uttar Pradesh
  - Janta Hospital, Varanasi, Uttar Pradesh
  - IPGMER & SSKM Hospital, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No
Plan to publish the findings after completion of the study.

REFERENCES:
- [Background] Lavhale MS, Havalad S, Gulati A. Resuscitative effect of centhaquin after hemorrhagic shock in rats. J Surg Res. 2013 Jan;179(1):115-24. doi: 10.1016/j.jss.2012.08.042. Epub 2012 Sep 2. PMID 22964270
- [Background] Geevarghese M 3rd, Patel K, Gulati A, Ranjan AK. Role of adrenergic receptors in shock. Front Physiol. 2023 Jan 16;14:1094591. doi: 10.3389/fphys.2023.1094591. eCollection 2023. PMID 36726848
- [Background] Papapanagiotou P, Xanthos T, Gulati A, Chalkias A, Papalois A, Kontouli Z, Alegakis A, Iacovidou N. Centhaquin improves survival in a swine model of hemorrhagic shock. J Surg Res. 2016 Jan;200(1):227-35. doi: 10.1016/j.jss.2015.06.056. Epub 2015 Jun 29. PMID 26216751
- [Background] Gulati A, Lavhale MS, Garcia DJ, Havalad S. Centhaquin improves resuscitative effect of hypertonic saline in hemorrhaged rats. J Surg Res. 2012 Nov;178(1):415-23. doi: 10.1016/j.jss.2012.02.005. Epub 2012 Apr 2. PMID 22487389
- [Background] Gulati A, Zhang Z, Murphy A, Lavhale MS. Efficacy of centhaquin as a small volume resuscitative agent in severely hemorrhaged rats. Am J Emerg Med. 2013 Sep;31(9):1315-21. doi: 10.1016/j.ajem.2013.05.032. Epub 2013 Jul 19. PMID 23871440
- [Background] Kontouli Z, Staikou C, Iacovidou N, Mamais I, Kouskouni E, Papalois A, Papapanagiotou P, Gulati A, Chalkias A, Xanthos T. Resuscitation with centhaquin and 6% hydroxyethyl starch 130/0.4 improves survival in a swine model of hemorrhagic shock: a randomized experimental study. Eur J Trauma Emerg Surg. 2019 Dec;45(6):1077-1085. doi: 10.1007/s00068-018-0980-1. Epub 2018 Jul 13. PMID 30006694
- [Background] Ranjan AK, Zhang Z, Briyal S, Gulati A. Centhaquine Restores Renal Blood Flow and Protects Tissue Damage After Hemorrhagic Shock and Renal Ischemia. Front Pharmacol. 2021 May 3;12:616253. doi: 10.3389/fphar.2021.616253. eCollection 2021. PMID 34012389
- [Background] Gulati A, Jain D, Agrawal NR, Rahate P, Choudhuri R, Das S, Dhibar DP, Prabhu M, Haveri S, Agarwal R, Lavhale MS. Resuscitative Effect of Centhaquine (Lyfaquin(R)) in Hypovolemic Shock Patients: A Randomized, Multicentric, Controlled Trial. Adv Ther. 2021 Jun;38(6):3223-3265. doi: 10.1007/s12325-021-01760-4. Epub 2021 May 10. PMID 33970455
- [Background] Gulati A, Choudhuri R, Gupta A, Singh S, Ali SKN, Sidhu GK, Haque PD, Rahate P, Bothra AR, Singh GP, Maheshwari S, Jeswani D, Haveri S, Agarwal A, Agrawal NR. A Multicentric, Randomized, Controlled Phase III Study of Centhaquine (Lyfaquin(R)) as a Resuscitative Agent in Hypovolemic Shock Patients. Drugs. 2021 Jun;81(9):1079-1100. doi: 10.1007/s40265-021-01547-5. Epub 2021 Jun 1. PMID 34061314
- [Derived] Khanna A, Vaidya K, Shah D, Ranjan AK, Gulati A. Centhaquine Increases Stroke Volume and Cardiac Output in Patients with Hypovolemic Shock. J Clin Med. 2024 Jun 27;13(13):3765. doi: 10.3390/jcm13133765. PMID 38999331